## **Study Protocol Cover Page**

**Document Title: Study Protocol** 

Study Official Title: Evaluation of Osteopathic Treatment in Adults with Nonspecific Neck

Pain

**NCT Number:** 

Date of Document: 12 November 2024

**Sponsor / Institution:** Istanbul Rumeli University

**Confidentiality Statement:** This document contains confidential information. Participants' names or personal identifiers are **not included**.

**Brief Description:** This study protocol describes a randomized, parallel-group interventional study comparing osteopathic treatment plus standard physical therapy versus standard physical therapy alone in adults with nonspecific neck pain. The protocol includes study objectives, eligibility criteria, interventions, outcome measures, and assessment schedule. The participants pain intensity (VAS), functional status (NDI), quality of life (SF-36), muscle strength, and cervical range of motion.

## **Statistical Cover Page**

**Document Title:** Statistical Analysis Plan

Study Official Title: Evaluation of Osteopathic Treatment in Adults with Nonspecific Neck

Pain

**NCT Number:** 

**Date of Document:** 12 November 2024

Sponsor / Institution: Istanbul Rumeli University

Confidentiality Statement: This document contains confidential information. Participants'

names or personal identifiers are not included.

**Brief Description:** The Statistical Analysis Plan outlines the methods for analyzing the primary and secondary outcomes of the study, including pain intensity (measured using the Visual Analog Scale, VAS), functional status (assessed using the Neck Disability Index, NDI), quality of life (evaluated using the Short Form-36, SF-36), muscle strength, and cervical range of motion. The plan describes statistical tests, significance thresholds, handling of missing data, and subgroup analyses for the randomized, parallel-group design. The Shapiro–Wilk test will be used to test the normality of data distribution. A paired sample t-test and an independent sample t-test will be used. A p-value of less than 0.05 (p < 0.05) will be considered statistically significant for all analyses.